CLINICAL TRIAL: NCT04814615
Title: A Diagnostic Study of CD38-Targeted ImmunoPET of Myeloma: Phase 2 Trial of Clinical Applications
Brief Title: A Diagnostic Study of CD38-Targeted ImmunoPET of Myeloma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoag Memorial Hospital Presbyterian (Other)
Responsible Party: Principal Investigator, Gary Ulaner, Director Molecular Imaging and Therapy, Hoag Memorial Hospital Presbyterian
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 177-20-CA
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; 89Zr-daratumumab; Dartumumab; PET/CT
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: Individual dose of 89Zr-DFO-daratumumab will be requested from Memorial Sloan Kettering Cancer Center and received at the Hoag Family Cancer Institute radiopharmacy for each individual 89Zr-DFO-daratumumab administration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CD38-positive multiple myeloma (Experimental): Patients with CD38 positive multiple myeloma with be enrolled. Patients will undergo pretreatment evaluation with standard of care diagnostic tests, as well as experimental 89Zr-daratumumab PET/CT. Patients will then undergo a course of standard of care therapy as defined by a medical oncologist. Following therapy, patients will repeat standard of care diagnostic tests, as well as experimental 89Zr-daratumumab PET/CT. Data analysis will be performed to evaluate 89Zr-daratumumab against standard of care diagnostic tests for the detection and localization of active disease before and after therapy.
  Interventions: Drug: 89Zr-daratumumab PET/CT

INTERVENTIONS:
Drug: 89Zr-daratumumab PET/CT — CD38-targeting imaging
  Other Names: CD38-targeted imaging

SUMMARY:
Evaluation of myeloma disease burden is currently suboptimal. This limits treatment planning and evaluation of residual disease following treatment. 89Zr-DFO-daratumumab is a novel immunoPET tracer, designed to detect CD38 on myeloma cells and allow visualization of myeloma in a PET scanner. A phase I study of 89Zr-DFO-daratumumab demonstrated safety and successful visualization of myeloma with 89Zr-DFO-daratumumab. This will be a phase II study of 89Zr-DFO-daratumumab to evaluate potential clinical applications of this novel imaging agent.

DETAILED DESCRIPTION:
This will be a phase II clinical trial to assess the potential clinical value of 89Zr-DFO-daratumumab immunoPET. 60 patients with multiple myeloma (MM) and a plan for daratumumab containing combination therapy will be enrolled. Prior to therapy, current standard of care (SoC), as well as a research 89Zr-DFO-daratumumab PET/CT, tests will be performed. Patients will then undergo standard of care therapy for myeloma as defined by a medical oncologist and SoC response assessments as defined by the International Myeloma Working Group (IMWG). Upon suspected complete response (CR) or completion of 12 cycles of therapy, a repeat research 89Zr-DFO-daratumumab PET/CT will be repeated and standard of care minimal residual disease (MRD) assessment will be performed. This design will determine how 89Zr-DFO-daratumumab immunoPET compares with current methods of measuring and localizing disease prior to therapy, if immunoPET can predict response to therapy, and how immunoPET compares with current methods of detecting MRD after therapy.

The therapy in this trial is standard of care. The research component is the addition of a novel immunoPET imaging test before and after standard of care therapy, to determine if the novel imaging test adds value over current measures of myeloma disease burden.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 21 years of age
2. Histologically/immunohistochemistry-confirmed CD38-positive multiple myeloma
3. At least one tumor lesion on CT, MRI, or FDG PET/CT within 90 days of protocol enrollment
4. ECOG performance status 0 to 2
5. Written informed consent obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study

Exclusion Criteria:

1. Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study.
2. Life expectancy < 12 months
3. Patients who cannot undergo PET/CT scanning because of weight limits. PET/CT scanners may not be able to function with patients over 450 pounds.
4. History of anaphylactic reaction to humanized or human antibodies.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
89Zr-daratumumab PET/CT for pre-treatment multiple myeloma imaging | up to 3 years
  89Zr-daratumumab PET/CT will be compared against standard of care laboratory and imaging measurements of multiple myeloma prior to therapy
89Zr-daratumumab PET/CT for post-treatment multiple myeloma imaging | up to 3 years
  89Zr-daratumumab PET/CT will be compared against standard of care laboratory and imaging measurements of multiple myeloma following therapy
Prediction of response to therapy | up to 3 years
  Determine if tumor uptake of 89Zr-daratumumab predicts response to therapy

CONTACTS AND LOCATIONS:
Overall Officials: Leila Andreas, MS, Study Director — Hoag Memorial Hospital Presbyterian
Locations (2):
- United States (2):
  - Hoag Memorial Hospital Presbyterian, Irvine, California
  - University of Miami, Miami, Florida

IPD SHARING:
Plan to Share IPD: No